CLINICAL TRIAL: NCT03997526
Title: Reapplix 3C Patch® System for the Treatment of Diabetic Foot Ulcers: A Medicare Claims Study
Brief Title: 3C Patch® Medicare Claims Study
Status: Terminated | Type: Observational
Why Stopped: CMS status changed - 3C Patch is now fully covered (NCD) - Medicare will no longer be collecting claims under CED
Sponsor: Reapplix (Other)
Responsible Party: Sponsor
Other Study IDs: REAPCEDUS01
Record Dates: First submitted 2019-06-21; First posted 2019-06-25 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Diabetic Foot Ulcer
Keywords: 3C Patch; Reapplix; LeucoPatch
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- 3C Patch treatment: Medicare beneficiaries with diabetes and hard-to-heal non-healing ulcers of the foot will receive usual care (i.e., care consistent with the IWGDF guidance on use of interventions to enhance the healing of chronic ulcers of the foot in diabetes) supplemented by the application of the 3C Patch (A platelet-rich plasma gel patch comprised of distinct fibrin, platelet, and leukocyte substantially parallel layers, prepared without the use of any added reagents through a two-step centrifugation process)
  Interventions: Device: 3C Patch

INTERVENTIONS:
Device: 3C Patch — A platelet-rich plasma gel patch comprised of distinct fibrin, platelet, and leukocyte substantially parallel layers, prepared without the use of any added reagents through a two-step centrifugation process

SUMMARY:
This prospective study will compare incidence rates of complete hard-to-heal diabetic foot ulcer healing in Medicare beneficiaries following application of the 3C Patch® plus usual care, tested against a historical control group of similar patients that received usual care during a randomized controlled trial.

DETAILED DESCRIPTION:
This is a prospective, observational, longitudinal, claims-based study with a historical control group. Data will be collected via claim forms and will be extracted directly from the Centers for Medicare & Medicaid Services (CMS) Medicare Research Identifiable Files (RIFs), which contain all medical claims for 100% of Medicare beneficiaries enrolled in the Medicare fee-for-service program. The study will be conducted in accordance with relevant guidelines of a central institutional review board (IRB), relevant informed consent regulations, and all other applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Medicare beneficiaries diagnosed with diabetic foot ulcer and receiving at least one treatment with the 3C Patch® System.
* Eligible ulcers will be hard-to-heal, meaning that the cross-sectional area will decrease by less than 50% during a four week period prior to the first application of the 3C Patch® (percentage change in cross-sectional area determined clinically by the treating physician by estimation at examination).
* Eligible ulcer's cross-sectional area will increase by less than 25% during a 4-week period prior to the first application of the 3C Patch® (percentage change determined clinically by treating physician by estimation at examination)
* The cross-sectional area of the index ulcer will be ≥50 and ≤1000 mm2 at the end of the 4 week period prior to the first application of the 3C Patch® (size determined clinically by the treating physician by estimation at examination).
* Participants will have the capacity to understand study procedures, and will be able to provide written informed consent.

Exclusion Criteria:

* Presence of sickle-cell anemia, hemophilia, thrombocytopenia (<100x109/L) or other clinically significant blood dyscrasia
* Known potential infectivity of blood products, including known HIV and hepatitis
* Patient in dialysis
* Clinical signs of infection of the index ulcer or reason to suspect that infection is present
* Revascularization procedure in the affected limb planned, or undertaken within the 4 weeks prior to the first application of the 3C Patch®
* Current treatment with cytotoxic drugs or with systemically administered glucocorticoids or other immunosuppressants
* Treatment of foot ulcers with growth factors, stem cells or equivalent preparation within the 8 weeks prior to the first application of the 3C Patch®
* The need for continued use of negative pressure wound therapy
* Likely inability to comply with the need for follow up visits because of planned activity
* Participation in another interventional clinical foot ulcer-healing trial within the 4 weeks prior to the first application of the 3C Patch®
* Prior enrollment in this study
* Judgement by the investigator that the patient does not have the capacity to understand the study procedures or provide written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Medicare beneficiaries diagnosed with diabetic foot ulcer
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
Complete healing | within 20 weeks of the first application of the 3C Patch.
  Rate (%) of complete healing of hard-to-heal diabetic foot ulcers in Medicare beneficiaries following application of the 3C Patch®.

SECONDARY OUTCOMES:
Number of 3C Patch® treatments administered | 20 weeks
  The number of 3C Patch® treatments administered within 20 weeks of initial application of the 3C Patch®.
Major amputation - target limb | 24 weeks
  The incidence of major (above ankle) amputation affecting the target limb by 24 weeks
Major amputation - contralateral limb | 24 weeks
  The incidence of major amputation affecting the contralateral limb by 24 weeks
Minor amputation - target limb | 24 weeks
  The incidence of minor (below ankle) amputation affecting the target limb by 24 weeks
Minor amputation - contralateral limb | 24 weeks
  The incidence of minor amputation affecting the contralateral limb by 24 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Mayo Clinic, Phoenix, Arizona
  - Natchitoches Regional Medical Center, Natchitoches, Louisiana
  - Opelousas General Hospital Wound Center, Opelousas, Louisiana
  - Southeast Wound Care and Hyperbaric Medical Center, Cape Girardeau, Missouri
  - Regional One Physician Specialists, Poplar Bluff, Missouri
  - UNC Chapel Hill, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Game F, Jeffcoate W, Tarnow L, Jacobsen JL, Whitham DJ, Harrison EF, Ellender SJ, Fitzsimmons D, Londahl M; LeucoPatch II trial team. LeucoPatch system for the management of hard-to-heal diabetic foot ulcers in the UK, Denmark, and Sweden: an observer-masked, randomised controlled trial. Lancet Diabetes Endocrinol. 2018 Nov;6(11):870-878. doi: 10.1016/S2213-8587(18)30240-7. Epub 2018 Sep 19. PMID 30243803
- [Background] Londahl M, Tarnow L, Karlsmark T, Lundquist R, Nielsen AM, Michelsen M, Nilsson A, Zakrzewski M, Jorgensen B. Use of an autologous leucocyte and platelet-rich fibrin patch on hard-to-heal DFUs: a pilot study. J Wound Care. 2015 Apr;24(4):172-4, 176-8. doi: 10.12968/jowc.2015.24.4.172. PMID 25853474